CLINICAL TRIAL: NCT02040727
Title: Communications of Muscle and Bone
Brief Title: Effect of Resistance Training on Musculoskeletal Endocrine Interactions
Acronym: COMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lynae J. Hanks, PhD. RD, Post-Doctoral Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: COMB
Record Dates: First submitted 2013-12-10; First posted 2014-01-20 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Musculoskeletal and Metabolic Crosstalk
Keywords: Myokines; Osteokines; Glucose homeostasis; Puberty
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Resistance Trained (Active Comparator): No Participation in Resistance Training
  Interventions: Behavioral: No Resistance Training
- Resistance Trained (Experimental): Participation in Resistance Training
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training — Supervised strength training 3 days per week for 24 weeks
  Arms: Resistance Trained
Behavioral: No Resistance Training — No supervised strength training throughout the study
  Arms: Non-Resistance Trained

SUMMARY:
This project will evaluate the impact of resistance training on the synthesis and release of hormones and growth factors from the musculoskeletal system and the extent to which the communicative capacity influences glucose homeostasis In turn, the contribution of glucose regulation on the musculoskeletal system will also be evaluated. This small study will serve as a pilot/feasibility study to define a protocol for implementation of a resistance training intervention in the pediatric population. To establish feasibility, this study population is limited to overweight African American boys ages 7-11 years.

In light of well-established accolades of resistance training, historical recommendations for avoidance among the pediatric population have deterred implementation of resistance training interventions in young adolescents. However, contemporary data indicating a profound benefit of resistance training to the skeletal system in pre-adolescents has led to the Academy of Sports Medicine, as well as various other pediatric health interest groups, to support supervised programs incorporating resistance training in young children, emphasizing large muscle and core strengthening. To date, such trials have not been conducted in the pediatric population

DETAILED DESCRIPTION:
Early adolescence (pre-puberty) is associated with many physiological changes with the intersection of metabolic pathways and body composition at the core. Lifestyle behaviors provide substantial influence and the rise of sedentary behavior particularly among this population can exert profound disruption. Metabolic dysfunction associated with limited activity and thus limited strain on the muscles and bones is associated with poor musculoskeletal health. Metabolic disturbance within the system during critical periods of development such as pre-puberty confers long-term health consequences.

Communication across systems is reliant upon various hormones which interact on the regulation of glucose homeostasis, bone metabolism, and muscle development. While it is well-established that bone and muscle growth are dependent upon fuel utilization, factors secreted by bone and muscle have been recently shown to play an interactive role in glucose homeostasis. Data derived primarily from animal models have demonstrated maintenance of physiological levels promote optimal growth and development, whereas these hormones appear to have adverse effects when levels are altered. While the data in animals is compelling, translation in humans has not been conducted.

Speculatively, impaired glucose homeostasis, much attributable to decreased strain on the musculoskeletal system, promotes impairments in physiological roles of these hormones. As a result, disordered development may be of consequence, such that the bones grow bigger yet have impaired quality, and delivery of fuel to muscle is compromised. Obesity-induced perturbations in metabolism and tissue partitioning may be an added stress to the system, impairing muscle function, power, performance and overall quality. Strategies that optimize the protective effects of the musculoskeletal system may be encompassed by forced stress on the system via resistance training, known to influence synthesis and release of hormones involved in fuel delivery and utilization by muscle and bone. The strategy proposed will target optimization of musculoskeletal health, promoting synthesis and release of musculoskeletal-derived signals providing protection on metabolic health at a critical period of development.

ELIGIBILITY:
Inclusion Criteria:

* overweight
* early pubertal boys (Tanner stage <3)
* ages 7-12 years
* self-identified as Non-Hispanic Black.

Exclusion Criteria:

* type 1 or 2 diabetes
* musculoskeletal disorders
* disturbances in glucose or lipid metabolism
* use of thyroid medication, diuretics, beta-blockers, or any medication that potentially could affect body composition, the lipid profile, insulin sensitivity, or blood pressure
* allergy to EMLA cream
* history of eating disorders, cancer, kidney disease, endocrinopathy, liver disease, heart disease, or thyroid disease
* medically determined not to be able to engage in resistance training

Ages: 7 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Fasting plasma FGF-23 concentration | 0,8,12,16, 24 weeks
  Fibroblast Growth Factor-23
Fasting serum osteocalcin concentration | 0, 8, 12, 16, 24 weeks
Fasting serum insulin concentration | 0, 8, 12, 16, 24 weeks
Fasting serum glucose concentration | 0, 8, 12, 16, 24 weeks

SECONDARY OUTCOMES:
Bone mineral content | 0, 12, 24 weeks
  by DXA
Muscle strength | 0, 8, 12, 16, 24 weeks
Muscle density | 0, 12, 24 weeks
  by pQCT
Bone stress-strain index | 0, 12, 24 weeks
  by pQCT

OTHER OUTCOMES:
Resting energy expenditure | 0, 12, 24 weeks
  by indirect calorimetry
Total fat mass | 0, 12, 24 weeks
  by DXA
Total lean mass | 0, 12, 24 weeks
  by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Orlando M Gutierrez, MD, MMSc, Study Director — University of Alabama at Birmingham; Lynae J Hanks, PhD, RD, Principal Investigator — University of Alabama at Birmingham; Krista Casazza, PhD, RD, Study Director — University of Alabama at Birmingham; Marcas Bamman, PhD, Study Director — University of Alabama at Birmingham; Ambika Ashraf, MD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Hanks LJ, Gutierrez OM, Ashraf AP, Casazza K. Bone Mineral Content as a Driver of Energy Expenditure in Prepubertal and Early Pubertal Boys. J Pediatr. 2015 Jun;166(6):1397-403. doi: 10.1016/j.jpeds.2015.02.054. Epub 2015 Apr 1. PMID 25841541